CLINICAL TRIAL: NCT00536289
Title: The Use of Blunt Needles Does Not Reduce Needlestick Injury During Obstetrical Laceration Repair
Brief Title: Blunt Needles do Not Reduce Needlestick Injuries to Doctors During Suturing After Child-Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MUSC HR # 10870
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2006-01

CONDITIONS: Needlestick Injuries
Keywords: Blunt needles; obstetric lacerations; Needlestick injuries; Needlestick injuries to physicians
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sharp needles
  Interventions: Device: Blunt needle
- 2 (Experimental): Blunt tipped needles
  Interventions: Device: Blunt needle

INTERVENTIONS:
Device: Blunt needle — Blunt tipped suture needle

SUMMARY:
The hypothesis for this study is that use of blunt tipped needles used during the repair of an episiotomy (tear in the vagina after childbirth) will result in fewer needlestick injuries to the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric laceration requiring suturing

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2005-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Holes in surgeons gloves | After surgical repair

SECONDARY OUTCOMES:
Surgeon satisfaction with the needle assignment | After the surgical repair

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sullivan, MD MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States